CLINICAL TRIAL: NCT02023944
Title: Maintaining Cognitive Health in Aging Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E1389-P
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Healthy People Programs
Keywords: Memory; Aging; Healthy People; Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): 12-week course on memory and aging, consists of psychoeducation and skills training
  Interventions: Other: Memory and Aging Course
- Control, No Intervention (No Intervention): No Intervention, considered "treatment as usual"

INTERVENTIONS:
Other: Memory and Aging Course — This is a 12-week course that will provide participants with an understanding of what normal and pathological aging processes look like. It will also provide participants with methods to maintain healthy lifestyles as they continue to grow older.
  Arms: Intervention

SUMMARY:
Interventions aimed at disseminating information about cognitive aging and lifestyle factors that contribute to successful cognitive aging, in addition to providing broad cognitive skills training, may improve the psychological wellness and day-to-day functioning of the aging Veteran population. This 12-week course aims to teach older Veterans (age 50+) about brain aging, lifestyle factors that contribute to successful aging, and techniques that can boost cognition in daily life.

DETAILED DESCRIPTION:
The proportion of Veterans over age 65 has risen from 11% to 26% from 1980 to 1990, and is estimated to rise to over 50% by 2030. Due to the growing number of older Veterans, health issues specific to the aging Veteran population is a primary concern for the Veterans Health Administration. Fear of developing dementia is common among older adults and minor memory lapses that were previously of little concern may be misinterpreted as signaling the beginning stages of dementia. Although normal cognitive aging is not the same as pathological aging, the impact of normal age-related changes warrants intervention since it can cause emotional distress and functional difficulties impacting occupational, recreational, and social pursuits and subjective cognitive impairment, defined as a noticed cognitive change without objective evidence of decline on neuropsychological testing may be the earliest precursor for dementia. While cognitive changes can be expected as we age, there is a growing body of literature demonstrating that modifiable lifestyle factors can influence functional ability and quality of life as one ages. In addition, cognitive training may result in improvements in cognition and functioning in older adults. Unfortunately, many older adults lack knowledge about cognitive aging and the factors that contribute to successful cognitive aging, which limits their ability to make changes that can improve the odds of successful cognitive aging. The need to disseminate information related to brain health has recently been recognized by key agencies involved in promoting the welfare of older adults, including the National Institutes of Neurological Disorders and Stroke, Mental Health, and Aging as well as the Centers for Disease Control and Prevention and the Alzheimer's Association. The current study builds upon previous work on cognitive intervention in older adults by investigating a multi-component intervention which includes psychoeducation about cognitive aging, presentation of lifestyle factors that contribute to successful cognitive aging, and broad cognitive skills training. Using a randomized controlled trial design, 72 Veterans will be assigned to either the intervention group (36) or a no treatment control group (36). Veterans will undergo baseline assessment, which will be used for comparison immediately following the intervention and at 3 and 6 month followup. Outcomes include knowledge of cognitive aging, measures of psychological wellness, and indicators of cognitive and functional ability.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 50 and older who are concerned about their memory.
* Veterans age 50 and older who want to learn about memory processes.

Exclusion Criteria:

Participants will be excluded if they display impairment on a cognitive screening measure, as determined using age and education corrected criteria with a minimum 90% specificity (using criteria: Schretlen, Testa, and Pearlson, 2010) as follows:

* Age Education MMSE Cut-off Specificity Sensitivity
* 51-55 / 26 or <
* 56-60 / 25 or <
* 61-65 / 25 or <
* 66-70 / 25 or <
* 71-75 / 23 or <
* 76-80 / 23 or <
* 86+ / 22 or <
* Or self or informant reported diagnosis of a brain disorder affecting cognition such as Alzheimer's disease, Mild Cognitive Impairment, Parkinson's disease, other dementia, stroke, or brain injury or diagnosis of a major mental illness such as major depression, schizophrenia, or bipolar disorder; active alcohol or substance abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen O'Connor, PsyD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hisnanick JJ. Changes over time in the ADL status of elderly US veterans. Age Ageing. 1994 Nov;23(6):505-11. doi: 10.1093/ageing/23.6.505. PMID 9231946
- [Result] Commissaris CJ, Ponds RW, Jolles J. Subjective forgetfulness in a normal Dutch population: possibilities for health education and other interventions. Patient Educ Couns. 1998 May;34(1):25-32. doi: 10.1016/s0738-3991(98)00040-8. PMID 9697554
- [Result] Royall DR, Palmer R, Chiodo LK, Polk MJ. Declining executive control in normal aging predicts change in functional status: the Freedom House Study. J Am Geriatr Soc. 2004 Mar;52(3):346-52. doi: 10.1111/j.1532-5415.2004.52104.x. PMID 14962147
- [Result] Royall DR, Palmer R, Chiodo LK, Polk MJ. Executive control mediates memory's association with change in instrumental activities of daily living: the Freedom House Study. J Am Geriatr Soc. 2005 Jan;53(1):11-7. doi: 10.1111/j.1532-5415.2005.53004.x. PMID 15667370
- [Result] Dodge HH, Kita Y, Takechi H, Hayakawa T, Ganguli M, Ueshima H. Healthy cognitive aging and leisure activities among the oldest old in Japan: Takashima study. J Gerontol A Biol Sci Med Sci. 2008 Nov;63(11):1193-200. doi: 10.1093/gerona/63.11.1193. PMID 19038834
- [Result] Reisberg B, Shulman MB, Torossian C, Leng L, Zhu W. Outcome over seven years of healthy adults with and without subjective cognitive impairment. Alzheimers Dement. 2010 Jan;6(1):11-24. doi: 10.1016/j.jalz.2009.10.002. PMID 20129317
- [Result] Depp C, Vahia IV, Jeste D. Successful aging: focus on cognitive and emotional health. Annu Rev Clin Psychol. 2010;6:527-50. doi: 10.1146/annurev.clinpsy.121208.131449. PMID 20192798
- [Result] La Rue A. Healthy brain aging: role of cognitive reserve, cognitive stimulation, and cognitive exercises. Clin Geriatr Med. 2010 Feb;26(1):99-111. doi: 10.1016/j.cger.2009.11.003. PMID 20176296
- [Result] Unverzagt FW, Smith DM, Rebok GW, Marsiske M, Morris JN, Jones R, Willis SL, Ball K, King JW, Koepke KM, Stoddard A, Tennstedt SL. The Indiana Alzheimer Disease Center's Symposium on Mild Cognitive Impairment. Cognitive training in older adults: lessons from the ACTIVE Study. Curr Alzheimer Res. 2009 Aug;6(4):375-83. doi: 10.2174/156720509788929345. PMID 19689237
- [Result] Papp KV, Walsh SJ, Snyder PJ. Immediate and delayed effects of cognitive interventions in healthy elderly: a review of current literature and future directions. Alzheimers Dement. 2009 Jan;5(1):50-60. doi: 10.1016/j.jalz.2008.10.008. PMID 19118809
- [Result] Lustig C, Shah P, Seidler R, Reuter-Lorenz PA. Aging, training, and the brain: a review and future directions. Neuropsychol Rev. 2009 Dec;19(4):504-22. doi: 10.1007/s11065-009-9119-9. Epub 2009 Oct 30. PMID 19876740
- [Result] Anderson LA, Day KL, Beard RL, Reed PS, Wu B. The public's perceptions about cognitive health and Alzheimer's disease among the U.S. population: a national review. Gerontologist. 2009 Jun;49 Suppl 1:S3-11. doi: 10.1093/geront/gnp088. PMID 19525214
- [Result] Hendrie HC, Albert MS, Butters MA, Gao S, Knopman DS, Launer LJ, Yaffe K, Cuthbert BN, Edwards E, Wagster MV. The NIH Cognitive and Emotional Health Project. Report of the Critical Evaluation Study Committee. Alzheimers Dement. 2006 Jan;2(1):12-32. doi: 10.1016/j.jalz.2005.11.004. PMID 19595852
- [Derived] O'Connor MK, Kraft ML, Daley R, Sugarman MA, Clark EL, Scoglio AAJ, Shirk SD. The Aging Well through Interaction and Scientific Education (AgeWISE) Program. Clin Gerontol. 2018 Oct-Dec;41(5):412-423. doi: 10.1080/07317115.2017.1387212. Epub 2017 Dec 8. PMID 29220623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was recruited, assigned to the control group, and then dropped out before the baseline due to dissatisfaction with group assignment.
Groups:
- Intervention: 12-week course on aging
  Memory and Aging Course: This is a 12-week course that will provide participants with an understanding of what normal and pathological aging processes look like. It will also provide participants with methods to maintain healthy lifestyles as they continue to grow older.
- Control, No Intervention: No Intervention; considered "treatment as usual"
Period: Overall Study
Arm/Group | Intervention | Control, No Intervention
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control, No Intervention | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 22 | 22 | 44
Age, Continuous [Mean (Full Range); unit: years] | 73.6 [66.7 to 80.5] | 73.6 [66.7 to 80.5] | 73.6 [66.7 to 80.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49
Memory Controllability Inventory [Mean (Standard Deviation); unit: units on a scale] — 12 item questionnaire used to measure perceived control over memory as one ages, minimum 0, maximum 12, higher scores indicate greater perceived control
  units on a scale | 65.2 (9.8) | 57.4 (10.4) | 60.7 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Memory Aging Questionnaire-Revised
Description: Measures laypersons' knowledge of memory changes in adulthood for research or educational purposes using true/false/"don't know" questions, with half of the questions pertaining to normal memory aging and the other half covering pathological memory deficits due to non-normative factors, such as dementia. Test-retest reliability and convergent and discriminant validity were established at adequate levels. Minimum value is 0, maximum value is 28, higher scores indicate better knowledge of memory aging.
Time Frame: Within 1 week of start of program
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control, No Intervention
Number analyzed (Participants) | 25 | 24
units on a scale | 19.8 (2.7) | 19.5 (3.6)

2. Secondary Outcome: Multifactorial Memory Questionnaire (MMQ)
Description: The MMQ is a measure constructed to reflect aspects of memory that are potentially amenable to clinical intervention. The scale consists of three subscales - memory contentment, memory ability, and memory strategy use. Higher scores indicate, respectively, greater contentment, ability, and strategy use. Minimum 0, maximum 80
Time Frame: Within 1 week of start of program
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: 12-week course on memory and aging
  Memory and Aging Course: This is a 12-week course that will provide participants with an understanding of what normal and pathological aging processes look like. It will also provide participants with methods to maintain healthy lifestyles as they continue to grow older.
Arm/Group | Intervention | Control, No Intervention
Number analyzed (Participants) | 25 | 24
units on a scale
  Memory Contentment | 46.7 (12.8) | 38.7 (15.2)
  Memory Ability | 52.6 (8.4) | 50.5 (11.4)
  Memory Strategy | 41.0 (8.7) | 36.5 (7.1)

ADVERSE EVENTS:
Time Frame: Through the duration of the study
Arm/Group | Intervention | Control, No Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02023944/Prot_SAP_000.pdf